CLINICAL TRIAL: NCT03156790
Title: A Clinical Phase II Trial to Describe Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of Spectrila® With the Pharmaceutical Active Ingredient Recombinant L-Asparaginase in Adult Subjects With Newly Diagnosed Acute B-Cell Lymphoblastic Leukaemia
Brief Title: PK, PD, Safety and Immunogenicity of Spectrila in Adults With Acute B-cell Lymphoblastic Leukaemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-Spectrila.1/ALL
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute B-Cell Lymphoblastic Leukaemia
Keywords: recombinant L-Asparaginase; Spectrila®; Lymphoblastic Leukaemia; BRALL 2014
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spectrila® (Experimental): recombinant L-Asparaginase
  Interventions: Drug: Spectrila®

INTERVENTIONS:
Drug: Spectrila® — 3 intravenous doses of 10 000 U/m² BSA each during induction phase I of the underlying BRALL 2014 treatment protocol on Days 21, 23 and 25. Additionally, the subjects (standard risk subjects only) will receive doses of 10 000 U/m² BSA each on Days 2, 4, 6, 9, 11 and 13 of the consolidation phase II, III and VI of BRALL 2014 treatment protocol.
  Other Names: recombinant L-Asparaginase

SUMMARY:
This is a non-controlled, single-arm, open-label clinical trial to describe the PK, PD, immunogenicity and safety of ASNase. All subjects enrolled will receive the IP recombinant ASNase (Spectrila®). Since Spectrila is already approved in the European Economic Area for first-line treatment of ALL patients of all age groups and showed similar efficacy and safety in comparison to Asparaginase medac no blinding or control groups are necessary. As underlying treatment protocol the BRALL 2014 treatment protocol will be used.

DETAILED DESCRIPTION:
The BRALL (Brazilian Acute Lymphocytic Leukaemia) treatment protocol was developed to standardise adult ALL treatment in Brazil since previously each centre used a different protocol. As in other treatment regimens of study groups, ASNase is an important component of ALL therapy. The rationale of the BRALL protocol was to use less myelotoxic drugs as daunorubicin, etoposide and cyclophosphamide and focus on more specific ALL directed therapies as asparaginase and methotrexate. The higher asparaginase dose regimen was chosen in BRALL 2014 to strengthen ASNase as major component of the treatment protocol while etoposide administration is reduced. Native ASNase is widely used and the data investigating non-inferiority, safety and tolerability of Asparaginase medac vs. Spectrila received a positive opinion from the European Medicines Agency (EMA). Nevertheless, data on efficacy and safety of Spectrila in adults are limited. Therefore, robust data on PK, pharmacodynamics (PD), safety and immunogenicity of Spectrila will be investigated in this trial in subjects with de novo ALL. The measurement of ASNase activity is considered to correlate with clinical effectiveness and therefore chosen as primary objective.

Subjects eligible for participation in this clinical trial will be treated with 3 intravenous doses of Spectrila of 10 000 U/m² BSA each during induction phase I of the underlying BRALL 2014 treatment protocol. Spectrila will be administered on Days 21, 23 and 25. Additionally, the subjects (standard risk subjects only) will receive doses of 10 000 U/m² BSA Spectrila each on Days 2, 4, 6, 9, 11 and 13 of the consolidation phase II, III and VI of BRALL 2014 treatment protocol. One final Analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with newly diagnosed pathologically confirmed acute B-cell lymphoblastic leukaemia
2. Female or male subjects between 18 and 55 years of age (inclusive)
3. Subjects eligible for treatment and treated according to the underlying treatment protocol BRALL 2014
4. Written informed consent given freely after the nature of the trial and disclosure of data has been explained to the subject
5. The subject shows no evidence of a current infection with SARS-CoV-2 (as diagnosed by thorax tomography or PCR test or test for anti-SARS-CoV-2 antibodies).
6. The subject expresses his/her understanding of the trial procedures and willingness to abide by them during the course of the trial
7. Female subjects of child-bearing potential must use a highly effective method of contraception (pearl index less than 1%) such as complete sexual abstinence, combined oral contraceptive, vaginal hormone ring, transdermal contraceptive patch, contraceptive implant or depot contraceptive injection in combination with a second method of contraception like a condom or a cervical cap/diaphragm with spermicide during the trial and for at least 7 months after Spectrila discontinuation.
8. Men should use effective contraceptive measures and be advised to not father a child while receiving ASNase. As a precautionary measure it is recommended to wait at least for 4 months after completion of treatment.

Exclusion Criteria:

1. Pre-treatment with any ASNase preparation
2. Hypersensitivity to the active substance, Escherichia coli- ASNase preparation or to any of the excipients
3. Pancreatitis at the time of treatment initiation or history of pancreatitis
4. Pre-existing known coagulopathy
5. Severe liver function impairment (bilirubin > three times the upper limit of normal [ULN]; transaminases > ten times ULN)
6. History of serious haemorrhage or serious thrombosis
7. Other current malignancies
8. Uncontrolled active infection
9. Evidence of infection with severe acute respiratory syndrome coronavirus typ 2 (SARS-CoV-2), the human immunodeficiency virus, hepatitis B or C, human T-lymphotropic virus type I and II, syphilis or Chagas disease (American trypanosomiasis)
10. Pregnancy as verified by a positive pregnancy test or nursing woman
11. Active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely
12. Evidence or suspicion that the subject might not comply with the requirements of the trial protocol.
13. Evidence or suspicion that the subject is unwilling or unable to understand the information given to him/her within the informed consent procedure
14. Any other factor which in the investigator's opinion is likely to compromise the subject's ability to participate in the trial
15. The subject is an employee or direct relative of an employee of the contract research organisation (CRO) involved in the trial, the trial site or medac.
16. The subject is imprisoned or is lawfully kept in an institution.
17. The subject has participated within 3 months before screening or plans to participate in a clinical trial (except the underlying treatment protocol BRALL 2014).
18. Previous participation in this clinical trial -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Asparaginase (ASNase) activity trough levels | Day 21 until Day 31
  Assessment of induction phase response, defined as subjects with asparaginase (ASNase) activity trough levels in serum ≥ 100 U/L in induction phase

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Simoes, MD, Principal Investigator — Ribeirão Medical School Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto
Locations (8):
- Brazil (8):
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte
  - Universidade Estadual de Campinas, Campinas
  - Hospital das Clínicas da UFG, Goiânia
  - Hospital Rio Grande Natal, Natal
  - Hospital de Clínicas Porto Alegre, Pôrto Alegre
  - Hospital das Clínicas São Paulo USP, Ribeirão Preto
  - INCA Instituto Nacional do Cancer, Rio de Janeiro
  - Hospital Estadual Mario Covas, Santo André

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's homepage — http://www.medac.de